CLINICAL TRIAL: NCT06872528
Title: Comparison of Epidural Analgesia With Intra-Articular Infiltration Analgesia for Postoperative Total Knee Arthroplasty Analgesia: A Prospective, Randomized Controlled Trial
Brief Title: Comparison of Epidural Analgesia With Intra-Articular Infiltration Analgesia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Namik Kemal University (Other)
Responsible Party: Principal Investigator, Ahmet Gültekin, Associate Professor, Namik Kemal University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NamikKU-AGultekin-2
Record Dates: First submitted 2025-02-24; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Epidural; Analgesia; Local Infiltration
Keywords: Ranawat; Epidural analgesia; Knee replacement surgery
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Analgesia provided only with epidural analgesia (Active Comparator)
  Interventions: Other: Recording the amount of medication and the number of complications according to observational follow-up
- Analgesia provided with epidural analgesia and local infiltration (Active Comparator)
  Interventions: Other: Recording the amount of medication and the number of complications according to observational follow-up

INTERVENTIONS:
Other: Recording the amount of medication and the number of complications according to observational follow-up — Observational monitoring of patients and recording data for 24 hours

SUMMARY:
The results of combining infiltrative analgesia applied by orthopedists with epidural analgesia applied by anesthesiologists after knee replacement surgery will be compared.

It aims to compare epidural analgesia with the maximum reduction of postoperative pain in patients, as well as in terms of both analgesic and complications.

The study will include patients who have undergone knee replacement surgery for six months. In the study, we will compare the results of painkillers applied to the patient from the waist or knee after the waist numbing anesthesia, which includes some of the routinely applied protocols of your knee replacement surgery. It is a condition that will be monitored after surgery. The study aims to reduce maximum pain with two painkiller methods applied in small amounts or together. No interventional application will be made to the patient who will undergo surgery other than routine application. After the surgery, you will be asked verbally about your pain level and side effects at certain hours after the surgery and the amount of painkillers used and the amount of painkillers will be determined according to the follow-up hours (1st, 2nd, 6th, 12th, 24th and 48th hours after the surgery). In addition to these, complications will also be monitored. The results of patients who can be fully followed up at the end of 6 months will be presented as a scientific study.

ELIGIBILITY:
Inclusion Criteria:

1. Age range 18-75
2. Those who underwent surgery with combined spinal anesthesia
3. Drugs administered with combined spinal anesthesia and intra-articular infiltration analgesia

Exclusion Criteria:

1. Those who do not want to participate in the study
2. Those who underwent surgery under general anesthesia
3. Patients outside the specified age range
4. Patients with inadequate follow-up results (patient, drug and device related)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-28 (Estimated); Primary Completion 2025-09-28 (Estimated); Study Completion 2025-09-28 (Estimated)

PRIMARY OUTCOMES:
Amount of local anesthetic used for epidural analgesia | 6 months
  Is there a statistical difference between the two groups? Monitoring the effect of local infiltration on the amount of epidural analgesic agent
Differences between the two groups in terms of complications and need for additional analgesia | 6 months
  The effect of epidural analgesia and infiltration analgesia on complications and additional analgesia needs in patients

REFERENCES:
- [Background] Berninger MT, Friederichs J, Leidinger W, Augat P, Buhren V, Fulghum C, Reng W. Effect of local infiltration analgesia, peripheral nerve blocks, general and spinal anesthesia on early functional recovery and pain control in total knee arthroplasty. BMC Musculoskelet Disord. 2018 Jul 18;19(1):232. doi: 10.1186/s12891-018-2154-z. PMID 30021587
- [Background] Liu X, Zhang H, Zhang H, Guo M, Gao Y, Du C. Local infiltration vs epidural analgesia for postoperative pain control after total knee or hip arthroplasty: A meta-analysis of randomized controlled trials. Medicine (Baltimore). 2020 Oct 30;99(44):e22674. doi: 10.1097/MD.0000000000022674. PMID 33126306